CLINICAL TRIAL: NCT00216541
Title: Randomised Study to Evaluate the Effect of Early Intervention to Treat Anemia With Epoetin Alfa Versus Standard Use on Hemoglobin Levels and the Incidence of Blood Transfusions in Cancer Patients Receiving Chemotherapy
Brief Title: A Study of the Safety and Effectiveness of Epoetin Alfa on Hemoglobin Levels and Blood Transfusions in Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag B.V. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR003541
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2010-06

CONDITIONS: Anemia; Neoplasms
Keywords: Anemia; cancer; transfusion; chemotherapy; hemoglobin; standard care; epoetin alfa; epoetin; erythropoietin
MeSH Terms: conditions — Anemia; Neoplasms | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to evaluate the effect of early treatment with epoetin alfa in addition to best standard of care on hemoglobin levels and the need for red blood cell transfusions in cancer patients receiving chemotherapy as compared to patients receiving standard epoetin alfa treatment and best standard of care.

DETAILED DESCRIPTION:
Cancer patients often experience anemia due to the disease itself, chemotherapy, or both. Quality of life is also affected, due in part to the tiredness associated with anemia. Previous studies with epoetin alfa have suggested that early intervention with epoetin alfa results in higher hemoglobin levels and lower incidence of red blood cell transfusions than are achieved with delayed intervention. This is a randomized, open-label, explorative, sequential study that evaluates the effects of early treatment with epoetin alfa to determine its impact on hemoglobin values and the need for red blood cell transfusions as well as the safety of epoetin alfa when used in the prevention of anemia during chemotherapy in adult patients with cancer. During their current course of chemotherapy, patients will receive either early treatment with epoetin alfa or standard treatment with epoetin alfa (epoetin alfa administered when hemoglobin is <=10 g/dL), in addition to best standard care. Best standard care during chemotherapy may include red blood cell transfusions, white cell growth factors, folic acid, and iron supplementation, as needed. Effectiveness will be determined by the number of patients who receive an allogenic blood transfusion during the study and the change in hemoglobin at 3 or 4 weeks, 8 or 9 weeks, and 12 weeks, and at the end of the treatment period. Safety evaluations (incidence of adverse events, abnormal clinical laboratory tests, and vital signs) will be performed throughout the study. The study hypothesis is that cancer patients receiving chemotherapy who receive early treatment with epoetin alfa will have higher hemoglobin levels and fewer red blood cell transfusions than cancer patients receiving chemotherapy who receive standard treatment with epoetin alfa. This study will be conducted in the Netherlands and will only enroll European patients and will be generally well-tolerated. Epoetin alfa injections (40,000 units) under skin once a week either within 7 days after start of first chemotherapy cycle or from day hemoglobin is <=10 g/dL. Patients will receive epoetin alfa during the current course of chemotherapy or up to 24 weeks. Dose may be adjusted.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of cancer and planned to receive chemotherapy in 1, 2, 3, or 4 weekly schedules for a minimum of 8 weeks
* have a hemoglobin level of >10 grams per deciliter and <= 12 grams per deciliter within 14 days before the start of the first on-study chemotherapy cycle
* Eastern Cooperative Oncology Group (scale used by researchers to represent the level of activity a patient is capable of) score of 0 (able to carry out all normal activity without restriction) to 2 (ambulatory and capable of all self-care but unable to carry out any work)
* life expectancy of >=6 months
* female subjects postmenopausal for at least 1 year, surgically sterile or practicing an effective method of birth control

Exclusion Criteria:

* Clinically significant or uncontrolled disease/dysfunction of any body system that is not due to cancer or chemotherapy, including uncontrolled or severe cardiovascular disease, recent (< 6 months) myocardial infarction, uncontrolled high blood pressure, congestive heart failure, or uncontrolled or unexplained history of seizures
* planned surgery expected to influence hemoglobin levels, within the first 8 or 9 weeks of study entry
* major illness or infection within 1 month of study entry
* highly increased risk of thrombotic or other vascular events
* androgen therapy within 2 months of study entry
* anemia due to factors other than cancer/chemotherapy (e.g., severe hemolysis, gastrointestinal bleeding, or myelodysplastic syndromes)
* blood transfusion within 14 days prior to study entry
* pregnant or lactating females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2003-08; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin from the start of the study to 3 or 4, 8 or 9, and 12 weeks, and at the end of the treatment period

SECONDARY OUTCOMES:
Number of patients who receive an allogenic blood transfusion during the study

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag B.V. Clinical Trial, Study Director — Janssen-Cilag B.V.

REFERENCES:
- [Result] Schouwink JH, Codrington H, Sleeboom HP, Kerkhofs LG, Wormhoudt LW. Prevention of anaemia by early intervention with once weekly epoetin alfa during chemotherapy. Eur J Cancer. 2008 Apr;44(6):819-29. doi: 10.1016/j.ejca.2008.02.017. Epub 2008 Mar 17. PMID 18343652
- See also: Treatment with Recombinant Epoetin Alfa Started Upfront: A Randomised study with Eprex (TREASURE) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=269&filename=CR003541_CSR.pdf